CLINICAL TRIAL: NCT00104728
Title: Pilot Neoadjuvant Study of ZD1839 (IRESSA®) as Single Agent Preoperative Therapy for Clinical Stage 1A and 1B (T1-2N0), II (T1-2N1, T3N0) and Selected IIIA (T3N1) Non-Small Cell Lung Cancer (NSCLC) With Molecular Correlates
Brief Title: Neoadjuvant IRESSA As Single Agent PreopTherapy for NSCLC With Molecular Correlates
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Early Stopping Rule: Would not meet interim analysis goal to proceed with enrollment
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-13922; IRUSIRES0256 (Other: AstraZeneca)
Record Dates: First submitted 2005-03-03; First posted 2005-03-04 (Estimated); Results first posted 2012-10-31 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-09

CONDITIONS: Lung Cancer
Keywords: stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IA non-small cell lung cancer; stage IB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neoadjuvant ZD1839 Preoperative Therapy (Experimental): The ZD1839 250-mg tablet will be taken once a day, every day about the same time. It can be taken with or without food.
  At the time of surgery, investigators will collect tissue from the participant's tumor once it has been removed. This tissue will be used to study the effect of ZD1839 on tumor growth.
  Interventions: Drug: ZD1839

INTERVENTIONS:
Drug: ZD1839
  Other Names: IRESSA®; gefitinib

SUMMARY:
RATIONALE: Gefitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving gefitinib before surgery may shrink the tumor so it can be removed.

PURPOSE: This phase II trial is studying how well gefitinib works in treating patients who are undergoing surgery for stage I, stage II, or stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the effects of neoadjuvant gefitinib on downstream signaling pathways, including Src-Stat3, PI3K/Akt, ERK activity, and Bcl-2 family members in patients with resectable stage I-IIIA non-small cell lung cancer.
* Determine the effects of this drug on cell cycle and apoptosis within the primary tumor, by measuring changes in pre- and post-treatment Ki-67, Mcm2, cleaved caspase-3, and ApoTag, in these patients.

Secondary

* Determine the clinical response rate in patients treated with this drug.
* Determine the pathological response rate, defined as > 95% necrosis or fibrosis in the pathological specimen, in patients treated with this drug.
* Determine the metabolic activity of this drug in these patients.
* Determine the safety, tolerability, and feasibility of this drug, in terms of toxicity and post-treatment resectability, in these patients.
* Correlate plasma and tumor concentrations of this drug with changes in post-treatment molecular markers in these patients.
* Identify a gene profile that predicts response to this drug in these patients.

OUTLINE: This is an open-label, pilot study.

Patients receive oral gefitinib once daily for 4 weeks in the absence of disease progression or unacceptable toxicity.

Within 3 days after completion of gefitinib, patients undergo restaging evaluation. Patients whose disease is still considered resectable proceed to surgery. Patients undergo thoracotomy with lobectomy or pneumonectomy OR sleeve resection. Patients also undergo mediastinal lymph node dissection. After surgical resection, treatment with gefitinib may continue off study at the discretion of the principal investigator.

After completion of study therapy, patients are followed at 30 days, every 4 months for 1 year, every 6 months for 1 year, and then annually thereafter.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study within 12.5 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed resectable non-small cell lung cancer (NSCLC), meeting 1 of the following clinical staging criteria:

  * Stage IA or IB (T1-2, N0)
  * Stage II (T1-2, N1 with negative mediastinoscopy or T3, N0)
  * Stage IIIA (T3, N1 with negative mediastinoscopy)

    * Level 10 hilar nodes may be positive provided mediastinoscopy is negative
* The following are not allowed (as evidenced by clinical staging criteria [CT scan, positron-emission tomography (PET) scan, or mediastinoscopy):

  * Positive N2 lymph nodes (ipsilateral/subcarinal mediastinal lymph nodes)
  * Positive N3 lymph nodes (contralateral mediastinal/hilar and supraclavicular/scalene lymph nodes)
  * T4 primary tumor (malignant pleural effusion or mediastinal invasion)
  * Symptomatic tumors (T3, N0-1) involving the superior sulcus (i.e., Pancoast tumors)
* Measurable disease by contrast-enhanced CT scan
* No metastatic disease (except peribronchial or hilar lymph node involvement [N1]) by fludeoxyglucose F 18 PET scan
* No malignant pleural effusion by preoperative evaluation

  * Pleural effusions visible only on CT scan that are not large enough for safe thoracentesis are allowed
  * No exudative effusions (even if cytologically negative), as evidenced by any of the following:

    * Ratio of pleural fluid protein to serum protein > 0.5
    * Ratio of pleural fluid lactic dehydrogenase (LDH) to serum LDH ≥ 0.6
    * Pleural fluid LDH > 200 IU/L
* No superior vena cava syndrome
* No spinal cord compression

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Eastern Cooperative Oncology Group (ECOG) 0-1

Life expectancy

* Not specified

Hematopoietic

* WBC ≥ 4,000/mm^3
* Absolute granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST or ALT ≤ 2 times ULN
* Alkaline phosphatase ≤ 2 times ULN

Renal

* Creatinine < 1.5 times ULN

Cardiovascular

* No uncontrolled ventricular arrhythmia
* No myocardial infarction within the past 3 months

Pulmonary

* Pre-resection FEV_1 > 2.0 L OR
* Predicted post-resection FEV_1 > 1.0 L
* No clinically active interstitial lung disease

  * Chronic stable asymptomatic radiographic changes allowed
* No post-obstructive pneumonia

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Willing to provide tumor biopsy pre- and post-gefitinib administration AND undergo PET scan
* No known severe hypersensitivity to study drug or any of its excipients
* No uncontrolled major seizure disorder
* No unstable or uncontrolled diabetes mellitus
* No serious infection requiring IV antibiotics
* No grade 3 neuropathy
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No other unstable or serious medical condition that would preclude study treatment or surgery
* No psychiatric disorder that would preclude giving informed consent
* No psychological, familial, sociological, or geographical condition that would preclude study compliance and follow up
* No other significant clinical disorder or laboratory finding that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior or concurrent systemic chemotherapy for NSCLC

Endocrine therapy

* Not specified

Radiotherapy

* No prior or concurrent radiotherapy for NSCLC

Surgery

* Recovered from prior oncologic or other major surgery
* At least 5 years since prior resection of lung disease
* No prior surgery for NSCLC
* No concurrent ophthalmic surgery

Other

* More than 30 days since prior non-approved or investigational drugs
* No other concurrent therapy for NSCLC
* No other concurrent investigational therapy
* No concurrent use of any of the following medications:

  * Phenytoin
  * Carbamazepine
  * Barbiturates (e.g., phenobarbital)
  * Rifampin
  * Hypericum perforatum (St. John's wort)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2004-10; Primary Completion 2008-05 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric B. Haura, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Neoadjuvant ZD1839 Preoperative Therapy: The ZD1839 250-mg tablet will be taken once a day, every day about the same time. It can be taken with or without food.
  At the time of surgery, investigators will collect tissue from the participant's tumor once it has been removed. This tissue will be used to study the effect of ZD1839 on tumor growth.
  ZD1839 :
Period: Overall Study
Arm/Group | Neoadjuvant ZD1839 Preoperative Therapy
Started | 42 (42 consented on study)
Completed | 23
Not Completed | 19
Not completed — screen failures | 19

BASELINE CHARACTERISTICS:
Arm/Group | Neoadjuvant ZD1839 Preoperative Therapy
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Objective Response Rate according to Response Evaluation Criteria In Solid Tumors (RECIST) criteria. Investigators planned to use this pilot study of neoadjuvant ZD1839 in patients with resectable NSCLC to specifically correlate molecular parameters to the primary clinical study endpoint clinical response assessed by CT response and PET scan response of the primary tumor.
Time Frame: 3 years
Arm/Group | Neoadjuvant ZD1839 Preoperative Therapy
Number analyzed (Participants) | 0

2. Secondary Outcome: Frequency of Toxicity Related to Study Treatment
Description: Review of adverse events utilizing Common Toxicity Criteria (CTC) V3. To estimate the safety, tolerability, and feasibility of preoperative ZD1839 in patients with resectable Stage IA/IB, II and selected IIIA NSCLC by evaluating toxicity and operability after preoperative ZD1839.
Time Frame: 3 years
Arm/Group | Neoadjuvant ZD1839 Preoperative Therapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Neoadjuvant ZD1839 Preoperative Therapy
Serious Adverse Events (participants affected / at risk) | 0/42
Other Adverse Events (participants affected / at risk) | 3/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neoadjuvant ZD1839 Preoperative Therapy (N=42)
Constipation - unlikely to be related (Gastrointestinal disorders) | 1 (1)
Nausea - unlikely to be related (Gastrointestinal disorders) | 1 (1)
Pain - Abdomen - NOS - unlikely to be related (General disorders) | 1 (1)
Pneumothorax - unrelated (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Supraventricular and nodal arrhythmia - Atrial fibrillation - unrelated (Cardiac disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Pilot study. At the time of interim analysis, the second early stopping rule was invoked for lack of activity (not enough responses to continue). Study closed to accrual 5/9/08.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes